CLINICAL TRIAL: NCT02533895
Title: Monocyte-derived Dendritic Cells Loaded With Tumour Cell Lysates for the Treatment of Refractory Solid Tumours of Childhood
Brief Title: Cancer Immune Therapy for the Treatment of Refractory Solid Tumours of Childhood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Activartis Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUVAC1
Record Dates: First submitted 2015-07-23; First posted 2015-08-27 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Childhood Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment with AV0113 (Experimental): 14 sarcoma and 7 non-sarcoma are treated with AV0113, an anti-tumour immune therapy with autologous DCs loaded with tumour cell lysates in order to establish the feasibility and safety of tumour vaccination.
  Peripheral blood mononuclear cells (MNCs) are obtained from patients by leukocyte apheresis. Monocytes enriched by density gradient centrifugation from MNCs will be used to generate immature DCs. These immature DCs will be loaded with autologous tumour cell lysates obtained by needle biopsy or surgery prior to tumour vaccination. The antigen loaded immature DCs will then receive a final maturation stimulus transmitted by exposure to lipopolysaccharide and interferon-gamma. Maturation enables DCs to present antigen with high efficiency to T-lymphocytes.
  Interventions: Biological: AV0113 DC-CIT; Other: Data evaluation
- Historic control (Other): In order to be able to compare the survival data of 14 sarcoma patients treated with AV0113, 42 historic control sarcoma patients from the data base of the Department of Orthopaedics, Medical University Vienna, that will be matched for disease, recurrences, relapses etc. will be included into this study.
  Interventions: Other: Data evaluation

INTERVENTIONS:
Biological: AV0113 DC-CIT — Mature loaded DCs will be injected intra-nodally into tumour free lymph nodes or subcutaneously close to tumour free lymph nodes at weekly intervals for at least 6 weeks.
  Arms: Treatment with AV0113
Other: Data evaluation — For obtaining a clearer picture of AV0113's utility in the treatment of bone and soft tissue sarcoma, a LT follow-up investigation of the 14 Sarcoma patients, which will be treated using the AV0113 DC-CIT technology, is planned, in order to gather first evidence for a potential LT effect of DC-CIT with AV0113.
  Furthermore, a comparison of the 14 sarcoma patients treated with AV0113 DC-CIT with a cohort of matched historic control patients that were treated using standard of care will be conducted. It is planned to analyse 42 control sarcoma patients that will be matched for disease, recurrences, relapses etc

SUMMARY:
This is an un-blinded Phase 1 study in which 21 patients suffering from solid advanced paediatric malignancies (14 sarcoma and 7 non-sarcoma patients) are treated with AV0113, an anti-tumour immune therapy with autologous Dendritic Cells (DCs) loaded with tumour cell lysates, in order to investigate its safety and feasibility.

For obtaining a clearer picture of AV0113's utility in the treatment of bone and soft tissue sarcoma, a long-term (LT) follow-up investigation of the 14 sarcoma patients, which will be treated using the AV0113 Dendritic Cell Cancer Immune Therapy (DC-CIT) technology is planned, in order to gather first evidence for a potential LT effect of DC-CIT with AV0113.

Furthermore, a comparison of the 14 sarcoma patients treated with AV0113 DC-CIT with a cohort of matched historic control patients that were treated using standard of care will be conducted. It is planned to analyse 42 historic control sarcoma patients that will be matched for disease, recurrences, relapses etc.

DETAILED DESCRIPTION:
In this phase I trial 21 paediatric patients with solid tumours of childhood (14 sarcoma and 7 non-sarcoma patients) that have exhausted all conventional treatment options are recruited for the treatment with AV0113.

Peripheral blood mononuclear cells (MNCs) will be obtained from patients by leukocyte apheresis. Monocytes enriched by density gradient centrifugation from MNCs will be used to generate immature DCs by cultivation in recombinant human interleukin-4 (IL-4) and granulocyte-macrophage colony-stimulating-factor (GM-CSF). These immature DCs will be loaded with autologous tumour cell lysates obtained by needle biopsy or surgery prior to tumour vaccination.The antigen loaded immature DCs will then receive a final maturation stimulus transmitted by exposure to lipopolysaccharide (LPS) and interferon-gamma (IFN-gamma). Maturation enables DCs to present antigen with high efficiency to T-lymphocytes. Subsequently, mature loaded DCs will be injected subcutaneously close to tumour free lymph nodes or intra-nodally into tumour free lymph nodes at weekly intervals for at least 6 weeks.

It is anticipated to establish the feasibility and safety of tumour vaccination in the described clinical setting and to find some clinical and/or experimental evidence for the induction of an anti-tumour immune response.

For obtaining a clearer picture of AV0113's utility in the treatment of bone and soft tissue sarcoma, a long-term (LT) follow-up investigation of the 14 Sarcoma patients, which will be treated using the AV0113 DC-CIT technology is planned, in order to gather first evidence for a potential LT effect of DC-CIT with AV0113.

Furthermore, a comparison of the 14 sarcoma patients treated with AV0113 DC-CIT with a cohort of matched historic control patients that were treated using standard of care will be conducted. It is planned to analyse 42 historic control sarcoma patients that will be matched for disease, recurrences, relapses etc.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the safety and feasibility testing of AV0113

* Male and female patients with a malignant neoplasia shall be eligible for this protocol provided they have no more "conventional" treatment options and have measurable disease. There is no age limit for participation in this study provided that the tumour is typical for the group of refractory solid neoplasias of childhood.
* Patients must not be HIV-positive.
* Patients must have primary tumour tissue or cells available at sufficient number to allow treatment according to the protocol.
* Patients or legal guardians must sign an informed consent indicating that they are aware this is a research study and have been told of its possible benefits and toxic side effects. Patients or their guardians will be given a copy of the consent form.

Inclusion criteria for patients included in the long-term follow up and comparison with historic controls

* Patients suffering from bone or soft tissue sarcoma that received treatment with AV0113 or are documented in the database of the Medical University Vienna's Department of Orthopaedics.
* At least one disease recurrence after first CR or worse disease condition (e.g.: never reached CR).
* Diagnosis between 1992-2003 and/or "inclusion time point" during the years 2000-2004.
* Availability of date of death or of confirmation that patient is still alive (for the currentness of confirmation that patients are still alive only the time span from 1 April 2014 to 1 April 2015 is accepted).
* Patients not older than 27 years at their ITP.

Exclusion Criteria:

Exclusion criteria for the safety and feasibility testing of AV0113

* Any of the inclusion criteria not met.
* Any condition which, in the investigator's opinion, may pose a risk to the patient or will interfere with the study objectives.

Exclusion criteria for patients included in the long-term follow up and comparison with historic controls

* Date of "inclusion time point" and death or confirmation that patient is still alive at time of evaluation not available.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2000-02; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Determination of the long-term effect of AV0113 by counting the total survival time in days measured from inclusion time point to death. | 15 years
  Total survival time of sarcoma patients, that underwent DC-CIT, measured from the "inclusion time point" (ITP) until death, independent of subsequent surgeries after DC-CIT.
  In the treatment group the inclusion time point (ITP) is defined as the day of surgery of the surgically treated relapse immediately before DC-CIT.
Comparison of total survival times in days of sarcoma patients treated with AV0113 with total survival times of a cohort of matched historic control patients. | 15 Years
  Total survival time of sarcoma patients, that underwent DC-CIT, measured from the "inclusion time point" (ITP) until death, independent of subsequent surgeries after DC-CIT; in comparison with the survival time of matched historical control patients measured from the ITP until death independent of subsequent surgeries.
  In the treatment group the ITP is defined as the day of surgery of the surgically treated relapse immediately before DC-CIT. In the control group the ITP is defined as the time of the surgery performed for the treatment of the xth relapse after which the matching patient of the treatment group received DC-CIT.
Comparison of the percentage of treatment patients still alive after 2 years with the percentage of matched historic control patients still alive after 2 years. | 2 years
  Percentage of sarcoma patients that underwent DC-CIT with AV0113, still alive after 2 years measured from the ITP independent of subsequent surgeries after DC-CIT; in comparison with the percentage of matched historical control patients still alive after 2 years measured from the ITP, independent of subsequent surgeries.
  In the treatment group the ITP is defined as the day of surgery of the surgically treated relapse immediately before DC-CIT. In the control group the ITP is defined as the time of the surgery performed for the treatment of the xth relapse after which the matching patient of the treatment group received DC-CIT.
Comparison of the percentage of treatment patients still alive after 5 years with the percentage of matched historic control patients still alive after 5 years. | 5 years
  Percentage of sarcoma patients that underwent DC-CIT with AV0113, still alive after 5 years measured from the ITP independent of subsequent surgeries after DC-CIT; in comparison with the percentage of matched historical control patients still alive after 5 years measured from the ITP, independent of subsequent surgeries.
  In the treatment group the ITP is defined as the day of surgery of the surgically treated relapse immediately before DC-CIT. In the control group the ITP is defined as the time of the surgery performed for the treatment of the xth relapse after which the matching patient of the treatment group received DC-CIT.
Comparison of the percentage of treatment patients still alive after 10 years with the percentage of matched historic control patients still alive after 10 years. | 10 years
  Percentage of sarcoma patients that underwent DC-CIT with AV0113, still alive after 10 years measured from the ITP independent of subsequent surgeries after DC-CIT; in comparison with the percentage of matched historical control patients still alive after 10 years measured from the ITP, independent of subsequent surgeries.
  In the treatment group the ITP is defined as the day of surgery of the surgically treated relapse immediately before DC-CIT. In the control group the ITP is defined as the time of the surgery performed for the treatment of the xth relapse after which the matching patient of the treatment group received DC-CIT.

SECONDARY OUTCOMES:
Number of treatment patients in which vaccination with AV0113 was feasible. | 4 years
  Establishment of the feasibility of anti-tumour immune therapy with autologous DCs loaded with tumour cell lysates for the treatment of patients suffering from solid advanced paediatric malignancies.
Number of serious adverse events in total and number of serious adverse events related to AV0113 vaccination. | 4 years
  Assessment of the qualitative and quantitative toxicity of DC based anti-tumour immune therapy.
Fraction of patients with immune response to vaccine antigens as measured by DTH testing. | 4 years
  In vivo evaluation of the vaccination efficiency by delayed-type hypersensitivity (DTH) testing.
Listings of in-vitro immunological variables with an association with survival as measured by Cox regression. | 4 years
  In vitro characterization of the anti-tumour immunity generated by the tumour vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Windhager, Dr., Study Director — Department of Orthopaedics, Medical University Vienna
Locations (2):
- Austria (2):
  - Department of Orthopaedics, Medical University Vienna, Vienna
  - St. Anna Children's Hospital, Vienna

REFERENCES:
- [Background] Bleyer WA. The impact of childhood cancer on the United States and the world. CA Cancer J Clin. 1990 Nov-Dec;40(6):355-67. doi: 10.3322/canjclin.40.6.355. No abstract available. PMID 2121321
- [Background] Cheung NK. Immunotherapy. Neuroblastoma as a model. Pediatr Clin North Am. 1991 Apr;38(2):425-41. doi: 10.1016/s0031-3955(16)38085-3. PMID 2006085
- [Background] Mayer P, Handgretinger R, Bruchelt G, Schaber B, Rassner G, Fierlbeck G. Activation of cellular cytotoxicity and complement-mediated lysis of melanoma and neuroblastoma cells in vitro by murine antiganglioside antibodies MB 3.6 and 14.G2a. Melanoma Res. 1994 Apr;4(2):101-6. doi: 10.1097/00008390-199404000-00004. PMID 8069095
- [Background] Cheung NK, Lazarus H, Miraldi FD, Abramowsky CR, Kallick S, Saarinen UM, Spitzer T, Strandjord SE, Coccia PF, Berger NA. Ganglioside GD2 specific monoclonal antibody 3F8: a phase I study in patients with neuroblastoma and malignant melanoma. J Clin Oncol. 1987 Sep;5(9):1430-40. doi: 10.1200/JCO.1987.5.9.1430. PMID 3625258
- [Background] Handgretinger R, Baader P, Dopfer R, Klingebiel T, Reuland P, Treuner J, Reisfeld RA, Niethammer D. A phase I study of neuroblastoma with the anti-ganglioside GD2 antibody 14.G2a. Cancer Immunol Immunother. 1992;35(3):199-204. doi: 10.1007/BF01756188. PMID 1638557
- [Background] Murray JL, Cunningham JE, Brewer H, Mujoo K, Zukiwski AA, Podoloff DA, Kasi LP, Bhadkamkar V, Fritsche HA, Benjamin RS, et al. Phase I trial of murine monoclonal antibody 14G2a administered by prolonged intravenous infusion in patients with neuroectodermal tumors. J Clin Oncol. 1994 Jan;12(1):184-93. doi: 10.1200/JCO.1994.12.1.184. PMID 8270976
- [Background] Khanna C, Anderson PM, Hasz DE, Katsanis E, Neville M, Klausner JS. Interleukin-2 liposome inhalation therapy is safe and effective for dogs with spontaneous pulmonary metastases. Cancer. 1997 Apr 1;79(7):1409-21. doi: 10.1002/(sici)1097-0142(19970401)79:73.0.co;2-3. PMID 9083164
- [Background] Sinkovics JG, Horvath JC. Vaccination against human cancers (review). Int J Oncol. 2000 Jan;16(1):81-96. doi: 10.3892/ijo.16.1.81. PMID 10601552
- [Background] Pardoll DM. Inducing autoimmune disease to treat cancer. Proc Natl Acad Sci U S A. 1999 May 11;96(10):5340-2. doi: 10.1073/pnas.96.10.5340. No abstract available. PMID 10318881
- [Background] Roskrow MA, Dilloo D, Suzuki N, Zhong W, Rooney CM, Brenner MK. Autoimmune disease induced by dendritic cell immunization against leukemia. Leuk Res. 1999 Jun;23(6):549-57. doi: 10.1016/s0145-2126(99)00045-4. PMID 10374848
- [Background] Darnell RB, DeAngelis LM. Regression of small-cell lung carcinoma in patients with paraneoplastic neuronal antibodies. Lancet. 1993 Jan 2;341(8836):21-2. doi: 10.1016/0140-6736(93)92485-c. PMID 8093269
- [Background] Darnell RB. Onconeural antigens and the paraneoplastic neurologic disorders: at the intersection of cancer, immunity, and the brain. Proc Natl Acad Sci U S A. 1996 May 14;93(10):4529-36. doi: 10.1073/pnas.93.10.4529. PMID 8643438
- [Background] Connolly AM, Pestronk A, Mehta S, Pranzatelli MR 3rd, Noetzel MJ. Serum autoantibodies in childhood opsoclonus-myoclonus syndrome: an analysis of antigenic targets in neural tissues. J Pediatr. 1997 Jun;130(6):878-84. doi: 10.1016/s0022-3476(97)70272-5. PMID 9202608
- [Background] Aichele P, Kyburz D, Ohashi PS, Odermatt B, Zinkernagel RM, Hengartner H, Pircher H. Peptide-induced T-cell tolerance to prevent autoimmune diabetes in a transgenic mouse model. Proc Natl Acad Sci U S A. 1994 Jan 18;91(2):444-8. doi: 10.1073/pnas.91.2.444. PMID 8290546
- [Background] Aichele P, Brduscha-Riem K, Zinkernagel RM, Hengartner H, Pircher H. T cell priming versus T cell tolerance induced by synthetic peptides. J Exp Med. 1995 Jul 1;182(1):261-6. doi: 10.1084/jem.182.1.261. PMID 7540654
- [Background] Takahashi H, Takeshita T, Morein B, Putney S, Germain RN, Berzofsky JA. Induction of CD8+ cytotoxic T cells by immunization with purified HIV-1 envelope protein in ISCOMs. Nature. 1990 Apr 26;344(6269):873-5. doi: 10.1038/344873a0. PMID 2184369
- [Background] Toes RE, Offringa R, Blom RJ, Melief CJ, Kast WM. Peptide vaccination can lead to enhanced tumor growth through specific T-cell tolerance induction. Proc Natl Acad Sci U S A. 1996 Jul 23;93(15):7855-60. doi: 10.1073/pnas.93.15.7855. PMID 8755566
- [Background] Toes RE, Blom RJ, Offringa R, Kast WM, Melief CJ. Enhanced tumor outgrowth after peptide vaccination. Functional deletion of tumor-specific CTL induced by peptide vaccination can lead to the inability to reject tumors. J Immunol. 1996 May 15;156(10):3911-8. PMID 8621930
- [Background] Medzhitov R, Janeway CA Jr. Decoding the patterns of self and nonself by the innate immune system. Science. 2002 Apr 12;296(5566):298-300. doi: 10.1126/science.1068883. PMID 11951031
- [Background] Langenkamp A, Messi M, Lanzavecchia A, Sallusto F. Kinetics of dendritic cell activation: impact on priming of TH1, TH2 and nonpolarized T cells. Nat Immunol. 2000 Oct;1(4):311-6. doi: 10.1038/79758. PMID 11017102
- [Background] Felzmann T, Huttner KG, Breuer SK, Wimmer D, Ressmann G, Wagner D, Paul P, Lehner M, Heitger A, Holter W. Semi-mature IL-12 secreting dendritic cells present exogenous antigen to trigger cytolytic immune responses. Cancer Immunol Immunother. 2005 Aug;54(8):769-80. doi: 10.1007/s00262-004-0637-2. Epub 2005 Jan 13. PMID 15647926
- [Background] Huttner KG, Breuer SK, Paul P, Majdic O, Heitger A, Felzmann T. Generation of potent anti-tumor immunity in mice by interleukin-12-secreting dendritic cells. Cancer Immunol Immunother. 2005 Jan;54(1):67-77. doi: 10.1007/s00262-004-0571-3. PMID 15693141
- [Background] Dohnal AM, Graffi S, Witt V, Eichstill C, Wagner D, Ul-Haq S, Wimmer D, Felzmann T. Comparative evaluation of techniques for the manufacturing of dendritic cell-based cancer vaccines. J Cell Mol Med. 2009 Jan;13(1):125-35. doi: 10.1111/j.1582-4934.2008.00304.x. Epub 2008 Mar 17. PMID 18363835
- [Background] Dohnal AM, Witt V, Hugel H, Holter W, Gadner H, Felzmann T. Phase I study of tumor Ag-loaded IL-12 secreting semi-mature DC for the treatment of pediatric cancer. Cytotherapy. 2007;9(8):755-70. doi: 10.1080/14653240701589221. Epub 2007 Oct 4. PMID 17917887
- [Background] Traxlmayr MW, Wesch D, Dohnal AM, Funovics P, Fischer MB, Kabelitz D, Felzmann T. Immune suppression by gammadelta T-cells as a potential regulatory mechanism after cancer vaccination with IL-12 secreting dendritic cells. J Immunother. 2010 Jan;33(1):40-52. doi: 10.1097/CJI.0b013e3181b51447. PMID 19952957
- [Background] Jonuleit H, Schmitt E, Schuler G, Knop J, Enk AH. Induction of interleukin 10-producing, nonproliferating CD4(+) T cells with regulatory properties by repetitive stimulation with allogeneic immature human dendritic cells. J Exp Med. 2000 Nov 6;192(9):1213-22. doi: 10.1084/jem.192.9.1213. PMID 11067871
- [Background] Munn DH, Sharma MD, Lee JR, Jhaver KG, Johnson TS, Keskin DB, Marshall B, Chandler P, Antonia SJ, Burgess R, Slingluff CL Jr, Mellor AL. Potential regulatory function of human dendritic cells expressing indoleamine 2,3-dioxygenase. Science. 2002 Sep 13;297(5588):1867-70. doi: 10.1126/science.1073514. PMID 12228717
- [Background] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Background] Jonuleit H, Kuhn U, Muller G, Steinbrink K, Paragnik L, Schmitt E, Knop J, Enk AH. Pro-inflammatory cytokines and prostaglandins induce maturation of potent immunostimulatory dendritic cells under fetal calf serum-free conditions. Eur J Immunol. 1997 Dec;27(12):3135-42. doi: 10.1002/eji.1830271209. PMID 9464798
- [Background] ESMO / European Sarcoma Network Working Group. Bone sarcomas: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2012 Oct;23 Suppl 7:vii100-9. doi: 10.1093/annonc/mds254. No abstract available. PMID 22997441
- [Background] Longhi A, Errani C, De Paolis M, Mercuri M, Bacci G. Primary bone osteosarcoma in the pediatric age: state of the art. Cancer Treat Rev. 2006 Oct;32(6):423-36. doi: 10.1016/j.ctrv.2006.05.005. Epub 2006 Jul 24. PMID 16860938
- [Background] Kempf-Bielack B, Bielack SS, Jurgens H, Branscheid D, Berdel WE, Exner GU, Gobel U, Helmke K, Jundt G, Kabisch H, Kevric M, Klingebiel T, Kotz R, Maas R, Schwarz R, Semik M, Treuner J, Zoubek A, Winkler K. Osteosarcoma relapse after combined modality therapy: an analysis of unselected patients in the Cooperative Osteosarcoma Study Group (COSS). J Clin Oncol. 2005 Jan 20;23(3):559-68. doi: 10.1200/JCO.2005.04.063. PMID 15659502
- [Background] Bielack SS, Kempf-Bielack B, Branscheid D, Carrle D, Friedel G, Helmke K, Kevric M, Jundt G, Kuhne T, Maas R, Schwarz R, Zoubek A, Jurgens H. Second and subsequent recurrences of osteosarcoma: presentation, treatment, and outcomes of 249 consecutive cooperative osteosarcoma study group patients. J Clin Oncol. 2009 Feb 1;27(4):557-65. doi: 10.1200/JCO.2008.16.2305. Epub 2008 Dec 15. PMID 19075282
- [Background] Leavey PJ, Mascarenhas L, Marina N, Chen Z, Krailo M, Miser J, Brown K, Tarbell N, Bernstein ML, Granowetter L, Gebhardt M, Grier HE; Children's Oncology Group. Prognostic factors for patients with Ewing sarcoma (EWS) at first recurrence following multi-modality therapy: A report from the Children's Oncology Group. Pediatr Blood Cancer. 2008 Sep;51(3):334-8. doi: 10.1002/pbc.21618. PMID 18506764
- [Background] Zagars GK, Ballo MT, Pisters PW, Pollock RE, Patel SR, Benjamin RS, Evans HL. Prognostic factors for patients with localized soft-tissue sarcoma treated with conservation surgery and radiation therapy: an analysis of 1225 patients. Cancer. 2003 May 15;97(10):2530-43. doi: 10.1002/cncr.11365. PMID 12733153